# Prevalence and incidence of multiple revisions following knee arthroplasty in Denmark 1998-2021: A nationwide population-based study

Study acronym: EMKAR

Study protocol version: Version 1.0 - 08/06/2023

Martin Lindberg-Larsen, co-supervisor, MD, PhD 4

SAP version number with date: Version 1.0 - 28/07/2023

| Author and statistical analyst: Julius Tetens Hald, MD <sup>1,2</sup> | |
|---|---|
| Signature and date: | 2023, Sept 5 |
| Senior biostatistician: Robin Christensen, BSc/MSc/PhD <sup>2,3</sup> | |
| Signature and date: | 2023, Sept 4. |
| Biostatistician: Sabrina Mai Nielsen, BSc, MSc, PhD <sup>2, 3</sup> | |
| Signature and date: Sai Mri Ni | 4th of September, 2023 |
| Chief investigator/clinical lead: Anders Odgaard, MD, DMSc, FRCS <sup>1, 5</sup> | |
| Signature and date: | 5 September 2023 |
| Other contributors: | |
| Michael Mørk Petersen, co-supervisor, MD, DMSc $^{\rm 1}$ | |

# Affiliations:

- 1. Department of Orthopaedic Surgery, Rigshospitalet, Copenhagen University Hospital, Denmark
- 2. Section for Biostatistics and Evidence-Based Research, The Parker Institute, Bispebjerg and Frederiksberg Hospital, Copenhagen, Denmark.
- 3. Research Unit of Rheumatology, Department of Clinical Research, University of Southern Denmark, Odense University Hospital, Odense, Denmark.
- 4. Orthopaedic research unit, Department of Orthopaedic surgery and traumatology, Odense University Hospital, Department of Clinical Research, Denmark.
- 5. Department of Clinical Medicine, University of Copenhagen, Copenhagen, Denmark

Background and rationale Knee arthroplasty is a common procedure performed worldwide to improve the quality of life for patients with degenerative knee conditions, trauma, and tumours. Complications can occur after knee arthroplasty, which may lead to a revision procedure, where at least one implant is exchanged, added, or removed. As the number of primary procedures in the world is increasing, so is the corresponding number of revisions. Some patients may require additional revision procedures, and some may end in a negative spiral of repeated revisions; We define three or more revisions on the same knee as being 'multiply revised'. The clinical impression of multiply revised patients is that the repeated occurrence of complications has significant impacts on the patients' quality of life including chronic pain, decreased independence, and increased morbidity. No study has yet investigated the incidence and prevalence of multiply revised knee arthroplasty patients stratified by previous revisions. To improve the care of multiply revised patients, epidemiological information is required which is the rationale of this study.

**Objectives** The aim of this observational study is to investigate the incidence and prevalence of multiply revised knee arthroplasty patients in all Danish patients with primary knee arthroplasty.

**Hypothesis** The number and burden of knee arthroplasty revision procedures and patients in Denmark has increased dramatically in the last 23 years.

Methods This is an observational study. Data will be collected from all primary and revision knee arthroplasties performed in Denmark from January 1st 1998 to 31st December 2021. Data will be acquired from two registers: The Danish Knee Arthroplasty Register (DKR), containing surgeon-reported data on primary and revision knee arthroplasties. In addition, data will be acquired from Landspatientregisteret, which contains all clinical data collected during any visit to a public or private healthcare facility in Denmark.

### PICOTS

**Population**: All Danish citizens who have received a primary knee arthroplasty at a Danish healthcare facility, from the 1<sup>st</sup> of January 1998 the to 31<sup>st</sup> of December 2021

Intervention/Exposure Multiple revision knee arthroplasties in the same knee

Comparator: None

*Outcome (primary):* Annual standardized prevalence and incidence of n-grade revisions following knee arthroplasty between 1998 and 2021 in Denmark.

*Time:* Retrospectively, from the 1st of January 1998 to the 31st of December 2021, i.e., up to 24 years follow-up.

Study design: Observational retrospective register study.

### **Further statistical details**

**Power considerations:** A sample size calculation has not been performed, as our sample will be determined solely by the actual number of eligible patients available from the registries.

*Framework:* This is an observational study aimed at reporting the prevalence and incidence of multiple revised knee arthroplasty patients in Denmark. No formal statistical testing will be performed.

Statistical interim analyses and stopping guidance: Not applicable.

*Timing of final analysis:* Access to all data has been acquired. The final analysis will be performed after the completion and acceptance of the SAP by all participants.

*Timing of outcome assessment:* (see next section). *Confidence intervals and P values:* Not applicable.

*Multiplicity:* No formal statistical testing will be performed.

Statistical software: R, version 4.3.0 (or newer).

# 2. TABULAR PRESENTATION OF TIMING OF OUTCOME MEASUREMENTS

| Registry | Observation period | Variables relevant for this study |
|---|---|---|
| The Danish Knee<br>Arthroplasty Register | January 1 <sup>st</sup> 1998 – 31 <sup>st</sup> December<br>2021 | ID-key (number) |
| Artinoplasty Register | 2021 | Date of surgery (date) |
| | | Code for implant type (number) |
| | | Revision performed (yes/no) |
| | | Revision of tibial component (yes/no) |
| | | Revision of femoral component (yes/no) |
| | | Laterality (left/right) |
| | | Sex (male/female) |
| | | Age (number) |
| | | Indication for primary procedure (number) |
| | | Performing institution (number) |
| | | Duration of procedure (minutes) |
| Landspatientregisteret | January 1 <sup>st</sup> 1998 – 31 <sup>st</sup> December<br>2021 | ID-key (number) |
| | 2021 | Date of surgery (date) |
| | | Code for procedure (number) |
| | | Laterality (left/right) |
| | | Sex (male/female) |
| | | Age (number) |
| | | Performing institution (number) |
| | | Year of death or emigration (date) |

### 3. ELABORATIONS ON OUTCOMES AND DATA

### Data management, The Danish Knee Arthroplasty Register:

<u>ID-key:</u> unique identification key specifying patient. This key is an anonymized ID key in encrypted integer format, and hence, is **not** equal to the CPR number of the participants.

Date of surgery: The date that the procedure took place. In character (date) format.

### Code for implant type

For the Danish knee arthroplasty register a set of codes are used to specify the inserted implant.

Primary procedures are defined as the following codes:

- 1 = TKA
- 2 = medial UKA
- 3= lateral UKA
- 4 = patellofemoral UKA
- 5+7 = rotating hinge-prosthesis
- 6 = Resection prosthesis
- 9 = Partial resurfacing
- 100 = Rotating hinge-prosthesis with condyle resection
- 104 = Resection or segmental prosthesis
- 105 = Hemicap
- 107 = Episealer
- 119 = tibiaprosthesis w. stem

### Revision procedure performed:

If the procedure is a revision it is marked with yes, otherwise it is marked with no.

# Definition of major revision:

A revision in DKR is defined as a major revision, if either the femoral or the tibial component has been revised. A procedure is marked as a major revision if either one of the variables "Revision of tibial component" and/or "revision of femoral component" are marked as yes.

# Definition of major and minor revision

Major and minor revisions are defined as the following implant types:

- 1 = TKA
- 2 = medial UKA
- 3= lateral UKA
- 4 = patellofemoral UKA
- 5+7 = rotating hinge-prosthesis
- 6 = Resection prosthesis
- 9 = Partial resurfacing
- 10 = articulated cement spacer
- 11 = fixated cement spacer
- 100 = Rotating hinge-prosthesis with condyle resection
- 103 = Removal of patella component
- 104 = Resection or segmental prosthesis
- 105 = Hemicap
- 107 = Episealer
- 108 = Other removal
- 109 = New liner
- 110 = New patella component
- 112 = Exchange of femoral component

- 117 = Removal of tibia component
- 119 = Insertion of stemmed tibia component
- 120 = Exchange of tibia component

Laterality: Code for specifying right/left knee. 1 = right, 2 = left

<u>Sex:</u> Specifying the sex of the patient. M = male, F = female

Age: Number specifying the age of the patient at the time of performed procedure

<u>Indication for primary procedure:</u> Code specifying the indication for performing the primary procedure. The codes are:

- 1 = Idiopathic knee osteoarthritis
- 2 = Secondary arthritis
- 3 = Sequelae after tibia condyle fracture
- 4 = Sequelae after femur condyle fracture
- 5 = sequelae after patella fracture
- 6 = Rheumatoid arthritis
- 7 = Sequelae after other arthritis
- 8 = Haemophilia
- 9 = Tumour primary
- 10 = Tumour metastasis

<u>Performing institution:</u> Code specifying the performing institution. The codes are classified as SHAK-codes, developed by "Sundhedsdatastyrelsen". (https://medinfo.dk/sks/brows.php)

<u>Duration of procedure</u>: Number specifying the duration of the performed procedure. Given as minutes.

### Data management, Landspatientregisteret:

<u>ID-key:</u> unique identification key specifying patient. This key is an anonymized ID key in character format, and hence, is **not** equal to the CPR-number of the participants.

Date of surgery: The date that the procedure took place. In character (date) format.

<u>Code for procedure:</u> NOMESCO procedure codes are used in Landspatientregisteret. KNGB\* codes specify primary procedures, whereas KNGC\* codes specify revision procedures.

### Definition of major revisions in Landspatientregisteret

Revision procedures are marked with KNGC\* codes. The following KNGC codes define a major revision:

KNGC01: Secondary insertion of proximal component of uncemented partial prosthesis in knee

KNGC02: Secondary insertion of distal component of uncemented partial prosthesis in knee

KNGC03: Secondary insertion of patellofemoral component of uncemented partial prosthesis in knee

KNGC04: Secondary insertion of multiple components of uncemented partial prosthesis in knee

KNGC11: Secondary insertion of proximal component of cemented partial prosthesis in knee

KNGC12: Secondary insertion of distal component of cemented partial prosthesis in knee

KNGC13: Secondary insertion of patellofemoral component of cemented partial prosthesis in knee

KNGC14: Secondary insertion of multiple components of cemented prosthesis in knee

KNGC19: Secondary insertion of cemented partial prosthesis in knee without specification

KNGC20: Secondary insertion of all components in uncemented total prosthesis in knee

KNGC21: Secondary insertion of proximal component in uncemented total prosthesis in knee

KNGC22: Secondary insertion of distal component in uncemented total prosthesis in knee

KNGC24: Secondary insertion of multiple components un uncemented total prosthesis in knee

KNGC29: Secondary insertion of uncemented total prosthesis in knee without specification

KNGC30: Secondary insertion of all components of hybrid total prosthesis in knee

KNGC31: Secondary insertion of proximal component of hybrid total prosthesis in knee

KNGC32: Secondary insertion of distal component of hybrid total prosthesis in knee

KNGC34: Secondary insertion of more than one component of hybrid total prosthesis in knee

KNGC39: Secondary insertion of hybrid total prosthesis in knee without specification

KNGC40: Secondary insertion of all components of cemented total prosthesis in knee

KNGC41: Secondary insertion of proximal component of cemented total prosthesis in knee

KNGC42: Secondary insertion of distal component of cemented total prosthesis in knee

KNGC44: Secondary insertion of multiple components of cemented total prosthesis in knee

KNGC49: Secondary insertion of cemented total prosthesis in knee without specification

KNGC99: Other secondary insertion of prosthesis in knee

### Definition of minor revisions in Landspatientregisteret

Minor revisions are defined as the KNGC codes listed here:

KNGC02A: Secondary insertion of only polyethylene liner in uncemented partial prosthesis in knee

KNGC09: Secondary insertion of uncemented partial prosthesis in knee without specification

KNGC1: Secondary insertion of cemented partial prosthesis in knee

KNGC12A: Secondary insertion of only polyethylene liner in cemented partial prosthesis in knee

KNGC22A: Secondary insertion of only polyethylene liner in uncemented total prosthesis in knee

KNGC23: Secondary insertion of patellofemoral component in uncemented total prosthesis in knee

KNGC32A: Secondary insertion of only polyethylene liner in hybrid total prosthesis in knee

KNGC33: Secondary insertion of patellofemoral component in hybrid total prosthesis in knee

KNGC42A: Secondary insertion of only polyethylene liner in hybrid total prosthesis in knee

KNGC43: Secondary insertion of patellofemoral component of cemented total prosthesis in knee

KNGC59: Secondary insertion of interpolated prosthesis in knee

KNGC59A: Insertion of spacer in knee in connection with revision

KNGC99A: Secondary insertion of patella component

KNGS49: Incision or revision with placement of medication in case of infection in knee joint

<u>Laterality:</u> Code for specifying right/left knee. TUL1 = right, TUL2 = left

<u>Sex:</u> Specifying the sex of the patient. M = male, F = female

Age: Number specifying the age of the patient at the time of the performed procedure

<u>Performing institution:</u> Code specifying the performing institution. The codes are classified as SHAK-codes, developed by "Sundhedsdatastyrelsen". (https://medinfo.dk/sks/brows.php)

<u>Year of death:</u> The year in which the patient has died. The patient will be marked as "ALIVE" if death has not occurred at the end of the observation period.

# Data management, for both registers.

<u>Definition of a revision:</u> A revision is defined as the exchange, addition, or removal of a knee prosthesis component (1). However, knee arthrodesis and amputation are not included in this study.

<u>Definition of major revision:</u> A major revision is defined as exchange of the femoral component and/or the tibial component with subgroups of tibial, femoral and all component exchange (2).

<u>Definition of minor revision:</u> A minor revision is defined as the exchange of polyethylene liner and/or addition or revision of the patella component. Insertion/removal/exchange of spacers are also included in this category (2).

<u>Population</u>: The population is defined as the number of alive citizens in the state of Denmark. Annual populations are defined as the population in Denmark on the 1<sup>st</sup> of January that year. Additional data for sex and age of the population is acquired. Data for the population is acquired from Danmarks Statistik (3).

<u>In case of disagreement between registers:</u> In cases of discrepancy between the two registers, Landspatientregisteret will overrule the Danish Knee arthroplasty register concerning following variables:

Laterality

Date of surgery

Gender

Age

Performing institution

In cases of discrepancy between the two registers, the Danish Knee arthroplasty register will overrule Landspatientregisteret concerning following variables:

Procedure code Revision of tibia Revision of femur Indication

<u>Calculation of standardized prevalence:</u> Annual standardized prevalence is calculated as the number of patients living with a n-grade revision during a given year as a proportion of the population in Denmark (the 1<sup>st</sup> of January that year) (3). The prevalence is then multiplicated by 100,000 for standardization. This is done for each level of revision, each year. E.g., the standardized prevalence for 1998 is calculated as:

$$Standardized\ prevalence, 1998 = \frac{Number\ of\ knees\ living\ in\ 1998\ with\ a\ n-grade\ revision}{Total\ population\ in\ Denmark\ in\ 1998}*100,000$$

The prevalence is only calculated for revisions performed between January 1st 1998 and December 31st 2021.

<u>Calculation of standardized incidence</u>: Annual standardized incidence is calculated as the number of new n-grade revisions performed as a proportion of the population in Denmark during a specific year. The population size of Denmark is defined as the population size at January 1<sup>st</sup> for that year (3). The incidence is then multiplicated by 100,000 for standardization. This is done for each level of revision, each year. E.g., the standardized incidence for 1998 is calculated as:

$$Standardized\ incidence, 1998 = \frac{\textit{Number of new } n - \textit{grade revisions in the population in 1998}}{\textit{Total population in Denmark in 1998}}*100,000$$

Missing data: We expect to encounter some missing data. All missing data will be described.

### **Data validation:**

All variables used in the analysis will be checked for obvious outliers and inconsistencies.

### Data template:

Based on this SAP, the statistical analyst will develop a tailored data template illustrating the data structure required for the statistical analyses.

# 4. PROTOCOL DEVIATIONS WITH BEARING ON THIS STATISTICAL ANALYSIS PLAN

The following details in this SAP represent deviations from the protocol.

| Header in the protocol | Change | Reason |
|---------------------------|--------|--------|
| (currently no deviations) | | |

# **5. OUTLINE**

The anticipated (predefined) outline of the manuscript is illustrated below.

# Figure 1. Flow diagram

Anticipated plot design, illustrating potential reasons for exclusion:



**Table 1.** Characteristics of primary knee arthroplasty procedures.

Characteristics Primary knee arthroplasties

Age, years

Females, n (%)

Implant type, n (%)

- TKA
- Medial UKA
- Lateral UKA
- Patellofemoral UKA
- Unspecified UKA
- Rotating hinge prosthesis
- Rotating hinge prosthesis with condyle resection
- Resection prosthesis
- Partial resurfacing
- Unspecified implant type (KNGB09, KNGB14, KNGB99)
- Isolated patella

### Region for the procedure, n (%)

- Northern Region of Denmark
- Middle Region of Denmark
- Southern Region of Denmark
- Zealand Region of Denmark
- Capital Region of Denmark
- Private hospitals
- Unknown

### Indication for the primary procedure, n (%)

- Idiopathic knee osteoarthritis
- Secondary knee osteoarthritis
- Sequelae following tibia condyle fracture
- Sequelae following femur condyle fracture
- Sequelae following patella fracture
- Rheumatoid arthritis
- Sequelae following other arthritis
- Haemophilia
- Primary bone tumour
- Metastatic bone tumour
- Unknown

Duration of the procedure, minutes

Values are means (SD) unless otherwise stated.

Abbreviations: TKA = total knee arthroplasty. UKA = unicompartmental knee arthroplasty

### Further statistical information related to table 1:

Data will be presented as mean with standard deviation (SD) when normally distributed or as median with interquartile range in case of skewed data. Dichotomous and categorical data will be presented in proportions. Normality of the data will be assessed using Q-Q plots, and histograms.

 Table 2. Annual occurrence of primary procedures and major n-grade revisions.

| Year | Primary procedures, | 1 <sup>st</sup> revision, n | 2 <sup>nd</sup> revision, n | <br>n grade revision, n | Maximal grade of revision performed* |
|---|---|---|---|---|---|
| 1998 | | | | | |
| 1999 | | | | | |
| 2000 | | | | | |
| 2001 | | | | | |
| 2002 | | | | | |
| 2003 | | | | | |
| 2004 | | | | | |
| 2005 | | | | | |
| 2006 | | | | | |
| 2007 | | | | | |
| 2008 | | | | | |
| 2009 | | | | | |
| 2010 | | | | | |
| 2011 | | | | | |
| 2012 | | | | | |
| 2013 | | | | | |
| 2014 | | | | | |
| 2015 | | | | | |
| 2016 | | | | | |
| 2017 | | | | | |
| 2018 | | | | | |
| 2019 | | | | | |
| 2020 | | | | | |
| 2021 | | | | | |

Only grades of revisions with occurrences >10 are shown
\*The maximal grade of revision performed is defined as the single greatest grade of revision performed that year

 Table 3: Annual occurrence of all n-grade revisions (including both major and minor revisions).

| Year | 1 <sup>st</sup> revision | 2 <sup>nd</sup> revision | <br>n grade revision | Maximal grade of revision performed* |
|---|---|---|---|---|
| 1998 | | | | |
| 1999 | | | | |
| 2000 | | | | |
| 2001 | | | | |
| 2002 | | | | |
| 2003 | | | | |
| 2004 | | | | |
| 2005 | | | | |
| 2006 | | | | |
| 2007 | | | | |
| 2008 | | | | |
| 2009 | | | | |
| 2010 | | | | |
| 2011 | | | | |
| 2012 | | | | |
| 2013 | | | | |
| 2014 | | | | |
| 2015 | | | | |
| 2016 | | | | |
| 2017 | | | | |
| 2018 | | | | |
| 2019 | | | | |
| 2020 | | | | |
| 2021 | | | | |

Only grades of revisions with occurrences >10 for all years are shown
\*The maximal grade of revision performed is defined as the single greatest grade of revision performed that year

Figure 2. The standardized prevalence and incidence rates of n-grade revisions from 1998 to 2021.

# Anticipated plot design, illustrating with imaginary data, A-D



Panel A and B illustrates standardized prevalence and incidence of <u>major</u> n-grade revisions. Panel C and D illustrate standardized prevalence and incidence of <u>all</u> n-grade revisions (including both major and minor revisions). Only grades of revisions with occurrences >10 are shown; for prevalence, >n-grade revisions are reported as well.

Figure 3. The standardized prevalence of patients with their total sum of revisions.



Panel A illustrates standardized prevalence of patients with major n-grade revisions. Panel B illustrates standardized prevalence rates of patients with all n-grade revisions (including major and minor revisions). The total sum of revisions is the summation of all revision procedures performed on a patient. E.g., a patient with 3 revisions performed on one knee and 4 revisions performed on the other knee, is categorized as a 7-grade revision patient. Only grades of revisions with occurrences >10 are shown as well as >n-grade grade revisions.

# SUPPLEMENTARY MATERIAL

The anticipated (predefined) supplementary material of the manuscript is illustrated below.

Supplementary file 1. Protocol

Supplementary file 2. This SAP

**Supplementary Figure 1.** Standardized annual prevalence (panel A) and incidence rates (panel B) for major n-grade revisions for male sex





**Supplementary Figure 2.** Standardized annual prevalence (panel A) and incidence rates (panel B) for major n-grade revisions for <u>female sex</u>.





**Supplementary Figure 3:** Standardized annual prevalence (panel A) and incidence rates (panel B) for major n-grade revisions for <u>age group 18-49.</u>





**Supplementary Figure 4:** Standardized annual prevalence (panel A) and incidence rates (panel B) for major n-grade revisions for <u>age group 50-69</u>.





**Supplementary Figure 5.** Standardized annual prevalence (panel A) and incidence rates (panel B) for major n-grade revisions for <u>age group 70-99.</u>





**Supplementary Figure 6:** Standardized annual prevalence (panel A) and incidence rates (panel B) for all n-grade revisions (including major and minor revisions) for <u>male sex</u>.





Only grades of revisions with occurrences >10 are shown; for prevalence, >n grade are reported as well.

**Supplementary Figure 7:** Standardized annual prevalence (panel A) and incidence rates (panel B) for all n-grade revisions (including major and minor revisions) for <u>female sex</u>.





Only grades of revisions with occurrences >10 are shown; for prevalence, >n grade are reported as well.

**Supplementary Figure 8:** Standardized annual prevalence (panel A) and incidence rates (panel B) for all n-grade revisions (including major and minor revisions) for <u>age group 18-49</u>.





**Supplementary Figure 9:** Standardized annual prevalence (panel A) and incidence rates (panel B) for all n-grade revisions (including major and minor revisions) for <u>age group 50-69.</u>





**Supplementary Figure 10:** Standardized annual prevalence (panel A) and incidence rates (panel B) for all n-grade revisions (including major and minor revisions) for <u>age group 70-99.</u>





**Supplementary table 1:** Age-stratified prevalence and incidence of major n-grade revisions for <u>females</u>, Denmark 2021.

| Grade of revision | Age group | No. of procedures | No. of persons in Denmark<br>on the 1 <sup>st</sup> of January in<br>2021 | Prevalence per 100.000 | Incidence per 100.000 |
|---|---|---|---|---|---|
| 1 <sup>st</sup> | Total | | | | |
| | 18-49 | | | | |
| | 50-69 | | | | |
| | 70-99 | | | | |
| 2 <sup>nd</sup> | Total | | | | |
| | 18-49 | | | | |
| | 50-69 | | | | |
| | 70-99 | | | | |
| 3 <sup>rd</sup> | Total | | | | |
| | 18-49 | | | | |
| | 50-69 | | | | |
| | 70-99 | | | | |
| 4 <sup>th</sup> | Total | | | | |
| | 18-49 | | | | |
| | 50-69 | | | | |
| | 70-99 | | | | |
| 5 <sup>th</sup> | Total | | | | |
| | 18-49 | | | | |
| | 50-69 | | | | |
| | 70-99 | | | | |
| n-grade | Total | | | | |
| | 18-49 | | | | |
| | 50-69 | | | | |
| | 70-99 | | | | |

**Supplementary table 2:** Age-stratified prevalence and incidence of major n-grade revisions for <u>males</u>, Denmark 2021.

| Grade of revision | Age group | No. of procedures | No. of persons in Denmark<br>on the 1 <sup>st</sup> of January in<br>2021 | Prevalence per 100.000 | Incidence per 100.000 |
|---|---|---|---|---|---|
| 1 <sup>st</sup> | Total | | | | |
| | 18-49 | | | | |
| | 50-69 | | | | |
| | 70-99 | | | | |
| 2 <sup>nd</sup> | Total | | | | |
| | 18-49 | | | | |
| | 50-69 | | | | |
| | 70-99 | | | | |
| 3 <sup>rd</sup> | Total | | | | |
| | 18-49 | | | | |
| | 50-69 | | | | |
| | 70-99 | | | | |
| 4 <sup>th</sup> | Total | | | | |
| | 18-49 | | | | |
| | 50-69 | | | | |
| | 70-99 | | | | |
| 5 <sup>th</sup> | Total | | | | |
| | 18-49 | | | | |
| | 50-69 | | | | |
| | 70-99 | | | | |
| n-grade | Total | | | | |
| | 18-49 | | | | |
| | 50-69 | | | | |
| | 70-99 | | | | |

**Supplementary table 3:** Age-stratified prevalence and incidence of all n-grade revisions (including major and minor revisions) for <u>females</u>, Denmark 2021

| Grade of revision | Age group | No. of procedures | No. of persons in Denmark<br>on the 1 <sup>st</sup> of January in<br>2021 | Prevalence per 100.000 | Incidence per 100.000 |
|---|---|---|---|---|---|
| 1 <sup>st</sup> | Total | | | | |
| | 18-49 | | | | |
| | 50-69 | | | | |
| | 70-99 | | | | |
| 2 <sup>nd</sup> | Total | | | | |
| | 18-49 | | | | |
| | 50-69 | | | | |
| | 70-99 | | | | |
| 3 <sup>rd</sup> | Total | | | | |
| | 18-49 | | | | |
| | 50-69 | | | | |
| | 70-99 | | | | |
| 4 <sup>th</sup> | Total | | | | |
| | 18-49 | | | | |
| | 50-69 | | | | |
| | 70-99 | | | | |
| 5 <sup>th</sup> | Total | | | | |
| | 18-49 | | | | |
| | 50-69 | | | | |
| | 70-99 | | | | |
| n-grade | Total | | | | |
| | 18-49 | | | | |
| | 50-69 | | | | |
| | 70-99 | | | | |

**Supplementary table 4:** Age-stratified prevalence and incidence of all n-grade revisions (including major and minor revisions) for <u>males</u>, Denmark 2021

| Grade of revision | Age group | No. of procedures | No. of persons in Denmark<br>on the 1 <sup>st</sup> of January in<br>2021 | Prevalence per 100.000 | Incidence per 100.000 |
|---|---|---|---|---|---|
| 1 <sup>st</sup> | Total | | | | |
| | 18-49 | | | | |
| | 50-69 | | | | |
| | 70-99 | | | | |
| 2 <sup>nd</sup> | Total | | | | |
| | 18-49 | | | | |
| | 50-69 | | | | |
| | 70-99 | | | | |
| 3 <sup>rd</sup> | Total | | | | |
| | 18-49 | | | | |
| | 50-69 | | | | |
| | 70-99 | | | | |
| 4 <sup>th</sup> | Total | | | | |
| | 18-49 | | | | |
| | 50-69 | | | | |
| | 70-99 | | | | |
| 5 <sup>th</sup> | Total | | | | |
| | 18-49 | | | | |
| | 50-69 | | | | |
| | 70-99 | | | | |
| n-grade | Total | | | | |
| | 18-49 | | | | |
| | 50-69 | | | | |
| | 70-99 | | | | |

# 6. REFERENCES

- 1. Price AJ, Alvand A, Troelsen A, Katz JN, Hooper G, Gray A, et al. Knee replacement. Lancet. 2018;392(10158):1672-82.
- 2. Klasan A, Magill P, Frampton C, Zhu M, Young SW. Factors predicting repeat revision and outcome after aseptic revision total knee arthroplasty: results from the New Zealand Joint Registry. Knee Surg Sports Traumatol Arthrosc. 2021;29(2):579-85.
- 3. Maradit Kremers H, Larson DR, Crowson CS, Kremers WK, Washington RE, Steiner CA, et al. Prevalence of Total Hip and Knee Replacement in the United States. J Bone Joint Surg Am. 2015;97(17):1386-97.
- 4. Gamble C, Krishan A, Stocken D, Lewis S, Juszczak E, Doré C, et al. Guidelines for the Content of Statistical Analysis Plans in Clinical Trials. Jama. 2017;318(23):2337-43.
- 5. Hiemstra B, Keus F, Wetterslev J, Gluud C, van der Horst ICC. DEBATE-statistical analysis plans for observational studies. BMC Med Res Methodol. 2019;19(1):233.

# 7. SAP REPORTING GUIDELINE

This SAP has been reported according to the items recommended by the DEBATE guideline for statistical analysis plans for observational studies (4, 5).

Table A. Recommended content of statistical analysis plans for observational studies

| ection/Item | Inde | X Description | Location in this SAP |
|---|---|---|---|
| ection 1: Administrative I | nform | nation | |
| Title and trial registration | 1a | Descriptive title that matches the protocol, with SAP either as a forerunner or subtitle, and study acronym | Front page |
| | 1b | Study registration number | - |
| SAP version | 2 | SAP version number with dates | Front page |
| Protocol version | 3 | Reference to version of protocol being used | Front page |
| SAP revisions | 4a | SAP revision history | Front page |
| | 4b | Justification for each SAP revision | Front page |
| | 4c | Timing of SAP revisions in relation to planned repetitive analyses | - |
| Roles and responsibility | 5 | Names, affiliations, and roles of SAP contributors | Front page |
| Signatures of: | 6a | Person writing the SAP | Front page |
| | 6b | Senior statistician responsible | Front page |
| | 6c | Chief investigator/clinical lead | Front page |
| Section 2: Introduction | | | |
| Background and rationale | 7 | Synopsis of study background and rationale including a brief description of research question and brief justification for undertaking the study | 1. Study overview |
| Objectives | 8 | Description of specific objectives and hypotheses, including secondary objectives | 1. Study overview |
| Section 3: Study Methods | | | • |
| Study design | 9 | Brief description of study design including type of study (e.g. case-control, cross-sectional or cohort study) | 1. Study overview |
| Power considerations | 10 | In case of an unspecified sample size, provide power calculations for (at least) the primary analysis or present a detectable difference with a specified power | 1. Study overview |
| Framework | 11 | Superiority, equivalence, or noninferiority hypothesis testing framework, including which comparisons will be presented on this basis | - |
| Statistical interim<br>analyses and stopping<br>guidance | 12a | Information on repetitive analyses specifying what repetitive analyses will be carried out and listing of time points | 1. Study overview |
| | 12b | Any planned adjustment of the significance level due to repetitive analyses | 1. Study overview |
| | 12c | Details of guidelines for stopping the study early | - |
| Timing of final analysis | 13 | Timing of final analysis, e.g., all outcomes analysed collectively or timing stratified by planned length of follow-up | 1. Study overview |
| Timing of outcome assessments | 14 | Time points at which the outcomes are measured including visit "windows" | 2. Tabular presentation of timing of outcome measurements |
| ection 4: Statistical Princi | ples | | |
| | 15 | Level of statistical significance | 1. Study overview |

| | | | - |
|---|---|---|---|
| Confidence intervals and | 16 | Description and rationale for any adjustment for multiplicity and, if so, detailing how the type 1 error is to be controlled | 1. Study overview |
| P values | 17 | Confidence intervals to be reported | 1. Study overview |
| Adherence and protocol deviations | 18a | Definition of protocol deviations for the study | 4. Protocol deviations with bearing on this statistical analysis plan |
| | 18b | Description of which protocol deviations will be summarized | 4. Protocol deviations<br>with bearing on this<br>statistical analysis plan |
| Analysis populations | 19 | Definition of analysis populations, eg, intention to treat, per protocol, complete case, safety | 5. Outline (for each table and figure) |
| Section 5: Study<br>Population | | | |
| Screening data | 20 | Reporting of screening data (if collected) to describe representativeness of trial sample | 5. Outline (Figure 1) |
| Eligibility | 21 | Summary of eligibility criteria | 1. Study overview |
| Recruitment | 22 | Information to be included in the STROBE flow diagram | 5. Outline (Figure 1) |
| Withdrawal/follow-up | 23a | Level of withdrawal, e.g., dropouts after inclusion or refusal to be contacted for additional information | 5. Outline (Figure 1) |
| | 23b | Timing of withdrawal/lost to follow-up data | 5. Outline (Figure 1) |
| | 23c | Reasons and details of how withdrawal/lost to follow-up data will be presented | 5. Outline (Figure 1) |
| Baseline patient characteristics | 24a | List of baseline characteristics to be summarized | 5. Outline (Table 1) |
| | 24b | Details of how baseline characteristics will be descriptively summarized | 5. Outline (Table 1) |
| Potential confounding covariates | 25 | A description of potential confounding covariates and how these will be dealt with | - |
| Section 6: Analysis | | | |
| Outcome definitions | | List and describe each primary and secondary outcome including details of: | |
| | 26a | Specification of outcomes and timings. If applicable include the order of importance of primary or key secondary endpoints (e.g., order in which they will be tested) | 5. Outline (mainly Table 2) |
| | 26b | Specific measurement and units (e.g., glucose control, HbA1c [mmol/mol or %]) | 5. Outline |
| | 26c | Any calculation or transformation used to derive the outcome (e.g., change from baseline, QoL score, time to event, logarithm, etc) | 5. Outline, and 3. Elaborations on outcomes and data |
| Analysis methods | 27a | What analysis method will be used and how the treatment effects will be presented | 5. Outline |
| | 27b | Any adjustment for covariates | 5. Outline |
| | 27c | Methods used for assumptions to be checked for statistical methods | 5. Outline |
| | 27d | Details of alternative methods to be used if distributional assumptions do not hold, eg, normality, proportional hazards, etc | 5. Outline |
| | 27e | Any planned sensitivity analyses for each outcome where applicable | 5. Outline |
| | 27f | Any planned subgroup analyses for each outcome including how subgroups are defined | 5. Outline |
| Missing data | 28 | Reporting and assumptions/statistical methods to handle missing data (e.g., multiple imputation) | 5. Outline |
| Additional analyses | 29 | Details of any additional statistical analyses required, eg, complier-average causal effect analysis | 5. Outline |
| Harms | 30 | Only applies when intervention effects are studied. Sufficient detail on summarizing safety data, e.g. information on severity, expectedness, and associations; details of how adverse events are scored; how adverse event data will be analysed and the follow-up time. | 5. Outline |
| Statistical software | 31 | Details of statistical packages to be used to carry out analyses | 1. Study overview |
| References | 22- | References to be provided for nonstandard statistical methods | 6. References |
| | 32a | References to be provided for floristandard statistical fliethods | o. Rejerences |
| | 32a<br>32b | Reference to Data Management Plan | - |

| 32c | Reference to the Study Master File and Statistical Master File | - |
|---|---|---|
| 32d | Reference to other standard operating procedures or documents to be adhered to | - |

Abbreviations: STROBE, STrengthening the Reporting of OBservational studies in Epidemiology; HbA1c, hemoglobin A1c; QoL, quality of life; SAP, statistical analysis plan.